CLINICAL TRIAL: NCT00351624
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effects of DHA on Cognitive Functions in Preschool Children
Brief Title: Effects of Docosahexaenoic Acid (DHA) on Cognitive Function in Children 4 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Martek #2006-1008
Record Dates: First submitted 2006-07-11; First posted 2006-07-13 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
Keywords: DHA supplementation; Cognitive function; Preschool children; Attention and behavior; Healthy Children
MeSH Terms: conditions — Behavior

ARMS (2):
- DHA (Active Comparator)
  Interventions: Behavioral: DHA
- placebo (Placebo Comparator)
  Interventions: Behavioral: placebo

INTERVENTIONS:
Behavioral: DHA
  Arms: DHA
Behavioral: placebo
  Arms: placebo

SUMMARY:
The primary objective of this study is to determine whether a 4-month period of supplementation with 400 mg/day of docosahexaenoic acid (DHA) provided from chewable softgel capsules containing bubblegum flavored microalgal oil (DHASCO-S) versus placebo improves one or more cognitive measures of attention, memory, processing speed, and error rate in healthy children 4 years of age.

The secondary objectives are to measure the safety and tolerability of the DHA dose administered and to measure blood DHA levels before and after supplementation.

DETAILED DESCRIPTION:
DHA is the primary omega-3 fatty acid present in the brain and retina and plays crucial structural and functional roles in these issues. The primary dietary source of DHA is fatty fish (e.g., salmon, herring, tuna). The American diet provides one of the lowest levels of omega-3 fatty acids of most industrialized nations. Children between the ages of 1 and 5 years consume only 30 to 50 mg DHA per day despite high requirements for this nutrient to support growth and tissue turnover.

Studies with human infants have reported visual and cognitive benefits of DHA supplementation in early life. Reported benefits include significant improvements on tests of visual acuity during infancy, psychomotor or mental development in the first two years of life, and problem-solving and sustained attention around 5 years of age.

Few studies have evaluated the effect that DHA supplementation has on the cognitive function of older children. Studies that considered DHA supplementation in children 4-12 years of age with attention-deficit/hyperactivity disorder (ADHD) or other developmental disorders have shown improvements on several measures of attention, behavior, and executive function.

Given the estimated high requirements of DHA to support growth and maintenance of the brain, the low consumption of DHA by American children, and the evidence from human and animal studies that DHA status affects the functional capacity of the central nervous system, there is a reasonable expectation that DHA supplementation administered to preschool-aged children will improve performance on tests of attention, memory, processing speed, and error rate.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age at enrollment between 4 years 0 months and 4 years 8 months
* Height and weight between the 10th and 90th percentiles of the National Center for Health Statistics (NCHS) growth charts
* Subject must meet normal developmental milestones.
* Subject able to understand instructions provided during the cognitive testing, i.e. English must be the primary language in the home
* No evidence of a medical condition that would preclude successful response or outcome (e.g., uncorrected vision or hearing impairment, attention deficit disorder, or inborn error of metabolism)
* Not taking any medications for seizure disorder, anxiety disorders (e.g., Valium or related compounds), ADHD (e.g., Ritalin, Adderall, Concerta, Strattera, or similar medication), childhood psychosis (e.g., Haldol, Risperdal), depression (e.g., Prozac), or for bipolar disorder. A subject will not be withdrawn from the trial if he/she needs to take one of these medications after enrollment. Antihistamines (e.g., Benadryl or other antihistamines) should not be administered within 24 hours of the day of the cognitive exams (Claritin or Allegra are allowed). If a subject is taking an antihistamine on the day of the cognitive tests, the tests will be rescheduled.

Exclusion Criteria:

* Premature birth (< 36 weeks gestation)
* Family history of ADHD
* Subject consumes > 3 oz. of fish more than 2 times per week.
* Subject consumes dietary supplements or foods containing or fortified with omega-3 fatty acids.
* Subject received any investigational product within the past 30 days.
* Subject having any medical condition that in the opinion of the principal investigator would preclude a successful response or outcome (e.g., uncorrected vision or hearing impairment, attention deficit disorder or inborn error of metabolism)

Ages: 4 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 216 (Actual)
Dates: Start 2006-05; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Leiter Test of Sustained Attention
Kiddie Continuous Performance Test (kCAP)
Peabody Picture Vocabulary Test
Day-Night Stroop Test

SECONDARY OUTCOMES:
Safety and tolerability of the DHA dose
Blood DHA levels before and after DHA supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Alan S Ryan, PhD, Study Director — DSM Nutritional Products, Inc.
Locations (10):
- United States (10):
  - Impact Clinical Trials, Los Angeles, California
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Northern Illinois Research Associates, DeKalb, Illinois
  - Pedia Research, Owensboro, Kentucky
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Eminence Research, LLC, Oklahoma City, Oklahoma
  - Prevention and Strengthening Solutions, Inc., Humboldt, Tennessee
  - Southwest Children's Research Associates, San Antonio, Texas
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Children's Hospital of the King's Daughters/Eastern Virginia Medical School, Norfolk, Virginia